CLINICAL TRIAL: NCT00406848
Title: Duloxetine Versus Placebo in the Long-Term Treatment of Patients With Late-Life Major Depression
Brief Title: A Study Comparing the Efficacy and Safety of Duloxetine and Placebo for the Treatment of Depression in Elderly Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10815; F1J-US-HMFA (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Results first posted 2010-09-29 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental)
  Interventions: Drug: duloxetine hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: duloxetine hydrochloride — Placebo for 1 week (double-blind placebo lead-in), then duloxetine 30 milligrams (mg) orally once daily (QD) for 1 week, followed by duloxetine 60 mg QD orally for 11 weeks. This double-blind acute treatment phase was followed by a double-blind 12 week continuation phase during which participants either remained on 60 mg QD or were eligible for dose escalation to 120 mg QD orally based on depression symptom severity.
  Other Names: LY248686, Cymbalta
  Arms: Duloxetine
Drug: placebo — Placebo for 13 weeks (The first week was placebo lead-in). This double-blind acute phase was followed by a double-blind 12 week continuation phase during which participants either remained on placebo or were eligible for receiving duloxetine 60 milligrams (mg) orally once daily (QD), beginning with duloxetine 30 mg QD orally for 1 week followed by duloxetine 60 mg QD orally for the remainder of the study based on depression symptom severity.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the efficacy and safety of duloxetine 60 mg once daily to placebo on depression in elderly patients (greater than or equal to 65 years of age). Patients who do not respond in the first 13 weeks will be eligible for rescue using pre-defined criteria. Patients randomized to duloxetine 60 mg/day meeting the rescue criteria will be increased to 120 mg/day. Patients randomized to the placebo arm meeting the rescue criteria will be assigned to duloxetine 60 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female outpatients at least 65 years of age who meet the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition Text Revision (DSM-IV-TR) diagnostic criteria for Major Depressive Disorder (MDD)
* Have a Mini Mental Score Exam (MMSE) score of at least 20 at Visit 1
* Have a degree of understanding such that the patient can communicate intelligibly with the investigator and study coordinator

Exclusion Criteria:

* Patients judged clinically to be at serious suicidal risk in the opinion of the investigator
* Have any prior history of bipolar disorder, panic disorder, psychosis, schizophrenia, or obsessive-compulsive disorder
* Have any current (within the past 12 months) DSM-IV-TR primary Axis I diagnosis other than MDD
* Have moderate to severe dementia
* Have a serious medical illness, including any cardiovascular (CV), hepatic, renal, respiratory, hematologic, endocrinologic, or neurologic disease, or clinically significant laboratory abnormality that is not stabilized or is anticipated to require hospitalization within 6 months, in the opinion of the investigator

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 370 (Actual)
Dates: Start 2006-11; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (33):
- United States (23):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pasadena, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherman Oaks, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamden, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coral Springs, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hoffman Estates, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Charles, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gaithersburg, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glen Burnie, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fall River, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olean, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lincoln, Rhode Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bartlett, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita Falls, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, West Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brown Deer, Wisconsin
- France (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arcachon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Douai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Limoges
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valence
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce, Puerto Rico

REFERENCES:
- [Derived] Harada E, Kato M, Fujikoshi S, Wohlreich MM, Berggren L, Tokuoka H. Changes in energy during treatment of depression: an analysis of duloxetine in double-blind placebo-controlled trials. Int J Clin Pract. 2015 Oct;69(10):1139-48. doi: 10.1111/ijcp.12658. Epub 2015 May 16. PMID 25980552
- [Derived] Nelson JC, Oakes TM, Liu P, Ahl J, Bangs ME, Raskin J, Perahia DG, Robinson MJ. Assessment of falls in older patients treated with duloxetine: a secondary analysis of a 24-week randomized, placebo-controlled trial. Prim Care Companion CNS Disord. 2013;15(1):PCC.12m01419. doi: 10.4088/PCC.12m01419. Epub 2012 Jan 3. PMID 23724353
- [Derived] Oakes TM, Katona C, Liu P, Robinson M, Raskin J, Greist JH. Safety and tolerability of duloxetine in elderly patients with major depressive disorder: a pooled analysis of two placebo-controlled studies. Int Clin Psychopharmacol. 2013 Jan;28(1):1-11. doi: 10.1097/YIC.0b013e32835b09cd. PMID 23138680
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study had a double-blind one-week placebo lead-in period before randomization, so baseline is defined as Week 1. 370 total patients were randomized and make up the safety analysis population. 299 of these patients were randomized under protocol amendments c, d and e, and make up the efficacy analysis population.
Groups:
- Duloxetine: Participants received placebo for 1 week (double-blind placebo lead-in) then started with duloxetine 30 milligrams (mg) orally once daily (QD) for 1 week, followed by duloxetine 60 mg QD orally for 11 weeks. This double-blind acute treatment phase was followed by a double-blind 12 week continuation phase during which participants either remained on 60 mg QD or were eligible for dose escalation to 120 mg QD orally based on depression symptom severity.
- Placebo: Participants received placebo for 13 weeks (The first week was placebo lead-in). This double-blind acute phase was followed by a double-blind 12 week continuation phase during which participants either remained on placebo or were eligible for receiving duloxetine 60 milligrams (mg) orally once daily (QD), beginning with duloxetine 30 mg QD orally for 1 week followed by duloxetine 60 mg QD orally for the remainder of the study based on depression symptom severity.
Period: Overall Study
Arm/Group | Duloxetine | Placebo
Started | 249 (Represents full safety analysis population. Efficacy analysis population (c,d,e) N=204.) | 121 (Represents full safety analysis population. Efficacy analysis population (c,d,e) N=95.)
Completed | 156 | 67
Not Completed | 93 | 54
Not completed — Withdrawal by Subject | 27 | 22
Not completed — Adverse Event | 38 | 7
Not completed — Lack of Efficacy | 9 | 14
Not completed — Protocol Violation | 10 | 6
Not completed — Lost to Follow-up | 6 | 2
Not completed — Physician Decision | 2 | 2
Not completed — Sponsor Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 249 | 121 | 370
Age Continuous [Mean (Standard Deviation); unit: years] | 72.89 (6.10) | 73.02 (5.64) | 72.93 (5.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 71 | 234
  Male | 86 | 50 | 136
Race/Ethnicity, Customized [Number; unit: Participants]
  African | 5 | 6 | 11
  Caucasian | 198 | 92 | 290
  Hispanic | 46 | 22 | 68
  Native American | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  France | 13 | 8 | 21
  United States | 195 | 94 | 289
  Mexico | 17 | 8 | 25
  Puerto Rico | 24 | 11 | 35
17 item Hamilton Depression Rating Scale Total Score(HAMD-17) [Mean (Standard Deviation); unit: units on a scale] — The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe). Results shown are based on efficacy analysis population only.
  units on a scale | 19.42 (5.56) | 19.32 (5.78) | 19.39 (5.62)
17 item Hamilton Depression Rating Scale (HAMD-17) - Maier subscale [Mean (Standard Deviation); unit: Units on a scale] — The Maier subscale (Items 1,2,7,8,9,10) represents symptoms of depression. Total subscale scores range from 0 (normal) to 24 (severe). Results shown are based on efficacy analysis population only.
  Units on a scale | 9.96 (3.11) | 10.08 (3.36) | 10.00 (3.19)
Geriatric Depression Scale (GDS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The 30-item Geriatric Depression Scale (GDS) is a self-administered test of 30 questions to measure the severity of depression. The yes/no questions result in a range of scores from 0 (normal) to 30 (severe depression). Results shown are based on efficacy analysis population only.
  units on a scale | 18.54 (6.91) | 17.64 (6.66) | 18.26 (6.83)
Numerical Rating Scale (NRS) Overall Pain Score [Mean (Standard Deviation); unit: units on a scale] — How much the participant has been bothered by pain over the last week, as measured by an 11-point Likert scale. A score of 0 reflects "not bothered at all" and a score of 10 reflects "extremely bothered". Results shown are based on efficacy analysis population only.
  units on a scale | 3.79 (2.96) | 3.59 (2.67) | 3.73 (2.87)
Brief Pain Inventory (BPI) 24-hour Average Pain Score [Mean (Standard Deviation); unit: units on a scale] — A self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). Results shown are based on efficacy analysis population only.
  units on a scale | 3.48 (2.70) | 3.48 (2.57) | 3.48 (2.66)
Mini Mental State Exam (MMSE) Total Score [Mean (Standard Deviation); unit: units on a scale] — Mini-Mental State Examination (MMSE)is a widely used rating measure of cognitive ability. The MMSE will be used to categorize patients as with or without dementia. Patients with a MMSE score of 20 to 23 will be categorized as having mild dementia, while those with a score of ≥ 24 will be categorized as having no dementia. Scores range from 0 to 30. Results shown are based on efficacy analysis population only.
  units on a scale | 28.55 (1.83) | 28.42 (1.72) | 28.51 (1.79)
Montgomery-Asberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Results shown are based on efficacy analysis population only.
  units on a scale | 29.25 (5.57) | 28.46 (5.40) | 29.00 (5.52)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 13 Weeks in Hamilton Depression Rating Scale (HAMD-17) Maier Subscale
Description: The Maier subscale (Items 1,2,7,8,9,10) represents symptoms of depression. Total subscale scores range from 0 (normal) to 24 (severe).
Time Frame: baseline (Week 1), Week 13
Population: All participants randomized under protocol amendment c,d,e, and have a baseline observation and at least one post-randomization observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 201 | 95
units on a scale | -4.34 (0.29) | -3.90 (0.44)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there would be no difference in changes from baseline (Week 1) to Week 13 on the HAMD-17 Maier subscale between duloxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.397, Mixed Models Analysis — The a priori threshold for statistical significance was 0.05; Mixed Model Repeated Measures (MMRM) analysis model: Change = Treatment + Pooled Investigator + Visit + Treatment* Visit + Baseline + Baseline*Visit

2. Secondary Outcome: Change From Baseline on the 30-item Geriatric Depression Scale (GDS)
Description: The 30-item Geriatric Depression Scale (GDS) is a self-administered test of 30 questions to measure the severity of depression. The yes/no questions result in a range of scores from 0 (normal) to 30 (severe depression).
Time Frame: baseline (Week 1), Week 13, Week 25
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 200 | 90
units on a scale
  Week 13 change | -6.01 (0.53) | -4.53 (0.79)
  Week 25 change | -7.02 (0.58) | -3.66 (1.00)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.115, Mixed Models Analysis — p-value is for difference between duloxetine and placebo on change from baseline (Week 1) to Week 13; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — p-value is for difference between duloxetine and placebo on change from baseline (Week 1) to Week 25; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in the HAMD-17 Total Score, Subscales, and Individual Items
Description: Total Score assess depression severity (scores 0-52). Core, Maier and Bech subscales assess symptoms of depression (scores:0-20=Core; 0-24=Maier; 0-22=Bech). Anxiety/Somatization subscale assesses severity of anxiety (0-18). Retardation subscale assesses dysfunction in mood and work (0-14). Sleep subscale assesses insomnia (0-6). Individual item scores may range from 0-4 or 0-2. Higher numbers indicate more severe symptoms.
Time Frame: baseline (Week 1), Week 13, Week 25
Population: Randomized patients with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 201 | 95
units on a scale
  Total - Week 13 Change | -7.42 (0.52) | -7.15 (0.77)
  Total - Week 25 Change | -8.98 (0.57) | -7.00 (1.01)
  Maier subscale Week 25 Change | -5.31 (0.29) | -4.17 (0.54)
  Bech subscale Week 13 Change | -4.35 (0.30) | -3.98 (0.46)
  Bech subscale Week 25 Change | -5.36 (0.31) | -4.07 (0.58)
  Core Mood subscale Week 13 Change | -3.29 (0.24) | -3.02 (0.36)
  Core Mood subscale Week 25 Change | -4.08 (0.23) | -3.00 (0.43)
  Anxiety/Somatization subscale Week 13 | -2.38 (0.20) | -2.26 (0.30)
  Anxiety/Somatization subscale Week 25 | -2.90 (0.22) | -2.44 (0.38)
  Sleep subscale Week 13 Change | -1.14 (0.12) | -1.14 (0.18)
  Sleep subscale Week 25 Change | -1.37 (0.13) | -1.35 (0.24)
  Retardation subscale Week 13 Change | -2.70 (0.21) | -2.73 (0.31)
  Retardation subscale Week 25 Change | -3.42 (0.20) | -2.77 (0.38)
  Item 1: Depressed Mood - Week 13 Change | -1.13 (0.09) | -1.02 (0.13)
  Item 1: Depressed Mood Week 25 Change | -1.36 (0.09) | -1.02 (0.16)
  Item 2: Feelings of Guilt Week 13 Change | -0.70 (0.06) | -0.60 (0.09)
  Item 2: Feelings of Guilt Week 25 Change | -0.91 (0.06) | -0.65 (0.12)
  Item 3: Suicide Week 13 Change | -0.16 (0.04) | -0.18 (0.05)
  Item 3: Suicide Week 25 Change | -0.19 (0.04) | -0.11 (0.07)
  Item 4: Insomnia Early Week 13 Change | -0.37 (0.06) | -0.29 (0.09)
  Item 4: Insomnia Early Week 25 Change | -0.42 (0.06) | -0.41 (0.12)
  Item 5: Insomnia Middle Week 13 Change | -0.40 (0.06) | -0.47 (0.09)
  Item 5: Insomnia Middle Week 25 Change | -0.49 (0.06) | -0.46 (0.11)
  Item 6: Insomnia Late Week 13 Change | -0.36 (0.06) | -0.41 (0.08)
  Item 6: Insomnia Late Week 25 Change | -0.45 (0.05) | -0.53 (0.10)
  Item 7: Work and Activities Week 13 Change | -0.82 (0.08) | -0.81 (0.12)
  Item 7: Work and Activities Week 25 Change | -1.12 (0.09) | -0.87 (0.16)
  Item 8: Retardation Week 13 Change | -0.48 (0.05) | -0.51 (0.08)
  Item 8: Retardation Week 25 Change | -0.57 (0.05) | -0.54 (0.09)
  Item 9: Agitation Week 13 Change | -0.39 (0.06) | -0.32 (0.08)
  Item 9: Agitation Week 25 Change | -0.45 (0.06) | -0.53 (0.11)
  Item 10: Anxiety/Psychic Week 13 Change | -0.81 (0.07) | -0.75 (0.11)
  Item 10: Anxiety/Psychic Week 25 Change | -0.98 (0.08) | -0.85 (0.14)
  Item 11: Anxiety (Somatic) Week 13 Change | -0.49 (0.06) | -0.55 (0.09)
  Item 11: Anxiety (Somatic) Week 25 Change | -0.70 (0.06) | -0.60 (0.11)
  Item 12: Somatic Symptom/Gastrointestinal Week 13 | -0.16 (0.04) | -0.20 (0.06)
  Item 12: Somatic Symptom/Gastrointestinal Week 25 | -0.23 (0.04) | -0.26 (0.07)
  Item 13: Somatic Symptoms/General Week 13 Change | -0.41 (0.06) | -0.40 (0.09)
  Item 13: Somatic Symptoms/General Week 25 Change | -0.52 (0.07) | -0.59 (0.13)
  Item 14: Genital Symptoms Week 13 Change | -0.29 (0.06) | -0.46 (0.08)
  Item 14: Genital Symptoms Week 25 Change | -0.41 (0.06) | -0.47 (0.12)
  Item 15: Hypochondriasis Week 13 Change | -0.47 (0.06) | -0.32 (0.08)
  Item 15: Hypochondriasis Week 25 Change | -0.49 (0.06) | -0.39 (0.11)
  Item 16: Loss of Weight Week 13 Change | -0.02 (0.03) | -0.09 (0.04)
  Item 16: Loss of Weight Week 25 Change | -0.13 (0.02) | -0.01 (0.04)
  Item 17: Insight Week 13 Change | -0.09 (0.02) | -0.10 (0.03)
  Item 17: Insight Week 25 Change | -0.07 (0.03) | -0.11 (0.05)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.773, Mixed Models Analysis — p-value is for HAMD-17 total score change from baseline (Week 1) to Week 13; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.084, Mixed Models Analysis — p-value is for HAMD-17 total score change from baseline (Week 1) to Week 25; Mixed Model Repeated Measures (MMRM) analysis model: Change =Treatment + Pooled Investigator + Visit + Treatment* Visit + Baseline + Baseline*Visit
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.059, Mixed Models Analysis — p-value is for Maier subscale change from baseline (Week 1) to Week 25; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.488, Mixed Models Analysis — p-value is for Bech subscale change from baseline (Week 1) to Week 13; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.048, Mixed Models Analysis — p-value is for HAMD-17 Bech subscale change from baseline (Week 1) to Week 25; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.529, Mixed Models Analysis — p-value is for Core Mood subscale change from baseline (Week 1) to Week 13; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.027, Mixed Models Analysis — p-value is for Core Mood subscale change from baseline (Week 1) to Week 25; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.749, Mixed Models Analysis — p-value is for Anxiety/Somatization subscale change from baseline (Week 1) to Week 13; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.296, Mixed Models Analysis — p-value is for Anxiety/Somatization subscale change from baseline (Week 1) to Week 25; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.984, Mixed Models Analysis — p-value is for Sleep subscale change from baseline (Week 1) to Week 13; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 11: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.930, Mixed Models Analysis — p-value is for Sleep subscale change from baseline (Week 1) to Week 25; Change = Treatment + Pooled Investigator + Visit + Treatment* Visit + Baseline + Baseline*Visit
Statistical Analysis 12: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.934, Mixed Models Analysis — p-value is for Retardation subscale change from baseline (Week 1) to Week 13; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 13: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.123, Mixed Models Analysis — p-value is for Retardation subscale change from baseline (Week 1) to Week 25; [statistical method as in outcome 3, analysis 2]

4. Secondary Outcome: Change From Baseline in the Brief Pain Inventory (BPI) Severity and Interference Scores
Description: The Brief Pain Inventory (severity and interference scales) (BPI) is a self-reported scale that measures the severity of pain and the interference of pain on function. Severity scores: 0 (no pain) to 10 (severe pain) on each question assessing worst pain, least pain, and average pain in past 24 hours, and pain right now. Interference scores: 0 (does not interfere) to 10 (completely interferes) on each question assessing interference of pain in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life.
Time Frame: baseline (Week 1), Week 13, Week 25
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 191 | 87
units on a scale
  Worst Pain - Week 13 | -0.66 (0.14) | -0.18 (0.19)
  Worst Pain - Week 25 | -0.74 (0.14) | -0.36 (0.20)
  Least Pain - Week 13 | -0.47 (0.11) | -0.00 (0.15)
  Least Pain - Week 25 | -0.54 (0.11) | -0.26 (0.16)
  Average Pain - Week 13 | -0.83 (0.13) | -0.14 (0.18)
  Average Pain - Week 25 | -0.87 (0.12) | -0.37 (0.18)
  Pain Right Now - Week 13 | -0.78 (0.13) | -0.26 (0.18)
  Pain Right Now - Week 25 | -0.86 (0.13) | -0.46 (0.18)
  Interference with General Activity - Week13 | -0.58 (0.13) | -0.03 (0.19)
  Interference with General Activity - Week 25 | -0.65 (0.13) | -0.23 (0.19)
  Interference with Mood - Week 13 | -0.82 (0.14) | -0.03 (0.19)
  Interference with Mood - Week 25 | -0.95 (0.13) | -0.25 (0.19)
  Interference with Walking Ability - Week 13 | -0.74 (0.14) | -0.19 (0.20)
  Interference with Walking Ability - Week 25 | -0.75 (0.15) | -0.24 (0.21)
  Interference with Normal Work - Week 13 | -0.72 (0.15) | -0.01 (0.21)
  Interference with Normal Work - Week 25 | -0.79 (0.15) | -0.19 (0.21)
  Int. with Relations with other people- Week 13 | -0.60 (0.13) | -0.03 (0.19)
  Int. with Relations with other people-Week 25 | -0.73 (0.13) | -0.18 (0.19)
  Interference with Sleep - Week 13 | -0.77 (0.15) | -0.17 (0.21)
  Interference with Sleep - Week 25 | -0.94 (0.14) | -0.26 (0.21)
  Interference with Enjoyment of Life- Week 13 | -0.93 (0.15) | 0.03 (0.21)
  Interference with Enjoyment of Life- Week 25 | -1.04 (0.15) | -0.08 (0.21)
  Average Interference Score - Week 13 | -0.76 (0.12) | -0.07 (0.17)
  Average Interference Score - Week 25 | -0.86 (0.12) | -0.19 (0.18)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.034, Mixed Models Analysis — p-value is for Severity of Worst Pain Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.100, Mixed Models Analysis — p-value is for Severity of Worst Pain - Week 25 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis — p-value is for Severity of Least Pain Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.126, Mixed Models Analysis — p-value is for Severity of Least Pain Week 25 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — p-value is for Severity of Average Pain Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis — p-value is for Severity of Average Pain Week 25 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.016, Mixed Models Analysis — p-value is for Severity of Pain Right Now Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.058, Mixed Models Analysis — p-value is for Severity of Pain Right Now Week 25 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis — p-value is for Interference with General Activity Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.060, Mixed Models Analysis — p-value is for Interference with General Activity Week 25 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 11: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — p-value is for Interference with Mood Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 12: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — p-value is for Interference with Mood Week 25 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 13: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis — p-value is for Interference with Walking Ability Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 14: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.040, Mixed Models Analysis — p-value is for Interference with Walking Ability Week 25 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 15: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — p-value is for Interference with Normal Work Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 16: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis — p-value is for Interference with Normal Work Week 25 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 17: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis — p-value is for Interference with Relations with Other People Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 18: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis — p-value is for Interference with Relations with Other People Week 25 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 19: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis — p-value is for Interference with Sleep Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 20: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — p-value is for Interference with Sleep Week 25 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 21: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — p-value is for Interference with Enjoyment of Life Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 22: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — p-value is for Interference with Enjoyment of Life Week 25 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 23: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — p-value is for Average Interference Score Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 24: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — p-value is for Average Interference Score Week 25 main effect of treatment; [statistical method as in outcome 3, analysis 2]

5. Secondary Outcome: Change From Baseline in the Numeric Rating Scales (NRS) for Pain Item Scores
Description: Numeric Rating Scales (Semantic Differential Scales) for Pain are 6 self-administered scales that assesses experience of overall pain, back pain, headache, shoulder pain, time in pain while awake, and pain interference with daily activities, during the past week. Each item is scored on a numeric 11-point semantic differential scale (0-10) from 0 = no pain to 10 = pain as severe as you can imagine; or 0 = none of the time to 10 = all of the time; or 0 = no interference to 10 = unable to do any activities at all.
Time Frame: baseline (Week 1), Week 13, Week 25
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 191 | 87
units on a scale
  Overall Pain - Week 13 | -0.65 (0.13) | -0.05 (0.18)
  Overall Pain - Week 25 | -0.67 (0.13) | -0.40 (0.19)
  Headaches - Week 13 | -0.32 (0.12) | 0.01 (0.16)
  Headaches - Week 25 | -0.28 (0.12) | 0.01 (0.18)
  Back Pain - Week 13 | -0.63 (0.14) | 0.00 (0.20)
  Back Pain - Week 25 | -0.75 (0.14) | -0.15 (0.21)
  Shoulder Pain - Week 13 | -0.54 (0.12) | -0.22 (0.17)
  Shoulder Pain - Week 25 | -0.55 (0.13) | -0.30 (0.18)
  Pain Interference with Daily Activities - Week 13 | -0.84 (0.14) | -0.20 (0.20)
  Pain Interference with Daily Activities - Week 25 | -0.91 (0.15) | -0.34 (0.21)
  Time in Pain While Awake - Week 13 | -0.75 (0.14) | -0.04 (0.19)
  Time in Pain While Awake - Week 25 | -0.80 (0.13) | -0.33 (0.20)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = .005, Mixed Models Analysis — p-value is for Overall Pain Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.204, Mixed Models Analysis — p-value is for Overall Pain Week 25 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.078, Mixed Models Analysis — p-value is for Headaches Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.147, Mixed Models Analysis — p-value is for Headaches Week 25 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis — p-value is for Back Pain Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis — p-value is for Back Pain Week 25 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.124, Mixed Models Analysis — p-value is for Shoulder Pain Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.231, Mixed Models Analysis — p-value is for Shoulder Pain Week 25 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis — p-value is for Interference with Daily Activities Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis — p-value is for Interference with Daily Activities Week 25 main effect of treatment; Change = Treatment + Pooled Investigator + Visit + Treatment* Visit + Baseline + Baseline*Visit
Statistical Analysis 11: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — p-value is for Time in Pain While Awake Week 13 main effect of treatment; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 12: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.036, Mixed Models Analysis — p-value is for Time in Pain While Awake Week 25 main effect of treatment; [statistical method as in outcome 3, analysis 2]

6. Secondary Outcome: Patient's Global Impression of Improvement (PGI-I) at 13 Weeks and 25 Weeks
Description: The PGI-Improvement scale is a patient-rated instrument that measures perceived improvement in symptoms. It is a 7-point scale where a score of 1 indicates that the patient is "very much improved," a score of 4 indicates that the patient has experienced "no change," and a score of 7 indicates that the patient is "very much worse."
Time Frame: Week 13, Week 25
Population: All participants randomized under protocol amendment c,d,e, and have at least one post-randomization observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 178 | 84
units on a scale
  Week 13 | 2.74 (0.13) | 3.02 (0.19)
  Week 25 | 2.38 (0.12) | 2.85 (0.23)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.214, Mixed Models Analysis — p-value is for PGI-I at Week 13; Mixed Model Repeated Measures (MMRM) analysis model: PGI-I = Treatment + Pooled Investigator + Visit + Treatment* Visit
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = .063, Mixed Models Analysis — p-value is for PGI-I at Week 25; Mixed Model Repeated Measures (MMRM) analysis model: PGI-I = Treatment + Pooled Investigator + Visit + Treatment* Visit

7. Secondary Outcome: Change From Baseline in the Clinical Global Impression-Severity (CGI-S)
Description: Measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: baseline (Week 1), Week 13, Week 25
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 203 | 94
units on a scale
  Week 13 Change | -1.25 (0.09) | -1.04 (0.13)
  Week 25 Change | -1.65 (0.09) | -1.17 (0.16)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = .162, Mixed Models Analysis — p-value is for change from baseline (Week 1) to Week 13; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = .009, Mixed Models Analysis — p-value is for change from baseline (Week 1) to Week 25; [statistical method as in outcome 3, analysis 2]

8. Secondary Outcome: Change From Baseline in the Mini-Mental State Exam (MMSE)
Description: Mini-Mental State Examination (MMSE)is a widely used rating measure of cognitive ability. Scores range from 0 to 30. The MMSE will be used to categorize patients as with or without dementia. Higher number indicates better cognitive ability. Patients with a MMSE score of 20 to 23 will be categorized as having mild dementia, while those with a score of ≥ 24 will be categorized as having no dementia.
Time Frame: baseline (Week 1), Week 9, Week 25
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 159 | 69
units on a scale
  Week 9 Change (n=159, n=69) | 0.12 (0.13) | 0.24 (0.18)
  Week 25 Change (n=161, n=71) | 0.29 (0.13) | 0.35 (0.18)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.555, ANCOVA — p-value is for change from baseline (Week 1) to Week 9; Model: Change = Treatment + Pooled Investigator + Baseline
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = .785, ANCOVA — p-value is for change from baseline (Week 1) to Week 25; Model: Change = Treatment + Pooled Investigator + Baseline

9. Secondary Outcome: Change From Baseline in the Quality of Life, Enjoyment, and Satisfaction Questionnaire (Q-LES-Q-SF)
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q-SF) measures the degree of enjoyment and satisfaction experienced in various areas of daily life. The short version is a self-administered 16 item scale evaluating satisfaction of general activities on a 5-point Likert scale that indicates the degree of enjoyment or satisfaction achieved during the past week (1 = very poor and 5 = very good).
Time Frame: baseline (Week 1), Week 13, Week 25
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 167 | 82
units on a scale
  Week 13 Change | 6.58 (0.71) | 5.27 (0.98)
  Week 25 Change (n=168, n=82) | 7.44 (0.78) | 4.79 (1.08)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.255, ANCOVA — p-value is for change from baseline (Week 1) to Week 13; Model: Change = Treatment + Pooled Investigator + Baseline
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.038, ANCOVA — p-value is for change from baseline (Week 1) to Week 25; Model: Change = Treatment + Pooled Investigator + Baseline

10. Secondary Outcome: Probability of Remission as Measured by the HAMD-17 Total Score ≤7 and ≤10
Description: Remission (visitwise binary outcome, yes/no) is defined as HAMD-17 Total Score ≤7 and ≤10. HAMD-17 measures depression severity. The total score can range from 0 (normal) to 52 (severe depression). The visitwise probability of patients meeting criteria for remission (either Total Score ≤7 or ≤10) was analyzed using a categorical, pseudo-likelihood-based repeated measures approach. This analysis included the fixed, categorical effects of treatment, investigator, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariate of baseline score.
Time Frame: Week 13, Week 25
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: probability of remission
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 201 | 95
probability of remission
  Remission (HAMD17 ≤ 7) - Week 13 | 0.37 (0.26) | 0.33 (0.42)
  Remission (HAMD17 ≤ 7) - Week 25 | 0.54 (0.22) | 0.49 (0.46)
  Remission (HAMD17 ≤ 10) - Week 13 | 0.54 (0.19) | 0.53 (0.31)
  Remission (HAMD17 ≤ 10) - Week 25 | 0.70 (0.21) | 0.72 (0.47)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.706, Mixed Models Analysis — p-values for Week 13 remission (HAMD17 ≤ 7); Mixed Model Repeated Measures (MMRM) analysis model: Remission = Treatment + Pooled Investigator + Visit + Baseline + Treatment*Visit
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.694, Mixed Models Analysis — p-values for Week 25 Remission HAMD17 ≤ 7; Mixed Model Repeated Measures (MMRM)analysis model:Remission = Treatment + Pooled Investigator + Visit + Baseline + Treatment*Visit
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.864, Mixed Models Analysis — p-values for Week 13 Remission - HAMD17 ≤ 10; [statistical method as in outcome 10, analysis 2]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.817, Mixed Models Analysis — p-values for Week 25 Remission - HAMD17 ≤ 10; [statistical method as in outcome 10, analysis 2]

11. Secondary Outcome: Probability of Response at Endpoint as Measured by ≥50% Improvement in the HAMD-17 Total Score
Description: Response (visitwise binary outcome, yes/no) is defined as ≥ 50% reduction from baseline in the HAMD-17 total score. HAMD-17 measures depression severity. The total score can range from 0 (normal) to 52 (severe depression). The visitwise probability of patients meeting criteria for response was analyzed using a categorical, pseudo-likelihood-based repeated measures approach. This analysis included the fixed, categorical effects of treatment, investigator, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariate of baseline score.
Time Frame: Week 13, Week 25
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: probability of response
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 201 | 95
probability of response
  Week 13 | 0.44 (0.19) | 0.48 (0.29)
  Week 25 | 0.61 (0.20) | 0.72 (0.46)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.664, Mixed Models Analysis — p-value is for probability of response at Week 13; Mixed Model Repeated Measures (MMRM)analysis model:Response = Treatment + Pooled Investigator + Visit + Baseline + Treatment*Visit
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.310, Mixed Models Analysis — p-value is for probability of response at Week 25; [statistical method as in outcome 11, analysis 1]

12. Secondary Outcome: Probability of Remission as Measured by the HAMD-17 Total Score ≤7 and ≤10 by Medical Comorbidity Severity as Assessed by the Cumulative Illness Rating Scale-Geriatric Version (CIRS-G)
Description: Remission defined as HAMD-17 Total Score ≤7 and ≤10. HAMD-17 measures depression severity. Total score ranges: 0 (normal) to 52 (severe depression). Visitwise probability of patients achieving remission was analyzed using a categorical, pseudo-likelihood-based repeated measures approach. CIRS-G evaluates 14 organ-specific categories using a rating strategy of 0=no problems; 1=current mild problem/past significant problem; 2=moderate disability/morbidity; 3=severe/constant significant disability; and 4=extremely severe/immediate treatment required/end organ failure. Total score ranges: 0 to 56.
Time Frame: Week 13, Week 25
Population: Randomized patients with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: probability of remission
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 201 | 95
probability of remission
  Remission HAMD-17 ≤ 7 Week 13 (CIRS-G ≥ 6) | 0.44 (0.07) | 0.44 (0.10)
  Remission HAMD-17 ≤ 7 Week 13 (CIRS-G < 6) | 0.33 (0.07) | 0.20 (0.10)
  Remission HAMD-17 ≤ 10 Week 13 (CIRS-G ≥ 6) | 0.53 (0.07) | 0.52 (0.10)
  Remission HAMD-17 ≤ 10 Week 13 (CIRS-G <6) | 0.53 (0.07) | 0.57 (0.14)
  Remission HAMD-17 ≤ 7 Week 25 (CIRS-G ≥ 6) | 0.52 (0.08) | 0.42 (0.13)
  Remission HAMD-17 ≤ 7 Week 25 (CIRS-G <6) | 0.53 (0.08) | 0.45 (0.25)
  Remission HAMD-17 ≤ 10 Week 25 (CIRS-G ≥ 6) | 0.71 (0.06) | 0.65 (0.12)
  Remission HAMD-17 ≤ 10 Week 25 (CIRS-G <6) | 0.63 (0.08) | 0.72 (0.25)

13. Secondary Outcome: Probability of Efficacy Onset as Measured by at Least 20% Sustained Reduction From Baseline in the HAMD-17 Maier Subscale at Week 3
Description: Patients are considered to have met onset (visitwise binary outcome, yes/no) criteria at a particular visit if they had at least 20% reduction from baseline in the HAMD-17 Maier subscale at that visit and at all subsequent visits in the acute phase. Maier subscale measures core symptoms of depression and scores range from 0 (normal) to 24 (severe). The visitwise probability of patients meeting onset criteria was analyzed using a categorical, pseudo-likelihood-based repeated measures approach.
Time Frame: Week 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Probability of onset
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 201 | 95
Probability of onset | 0.43 (0.04) | 0.30 (0.05)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.036, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM)analysis model: Onset = Treatment + Visit + Baseline + Treatment*Visit

14. Secondary Outcome: Change From Baseline in Supine Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Time Frame: baseline (Week 1), Week 13, Week 25
Population: All randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 246 | 118
mmHg
  Systolic BP Week 13 Change | 0.19 (0.94) | -0.58 (1.39)
  Diastolic BP Week 13 Change | 1.89 (0.62) | -1.58 (0.92)
  Systolic BP Week 25 Change | 2.22 (1.09) | 0.54 (1.99)
  Diastolic BP Week 25 Change | 2.44 (0.68) | 0.65 (1.23)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.637, Mixed Models Analysis — p-value is for Systolic BP change from baseline (Week 1) to Week 13; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — p-value is for Diastolic BP change from baseline (Week 1) to Week 13; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.452, Mixed Models Analysis — p-value is for Systolic BP change from baseline (Week 1) to Week 25; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.193, Mixed Models Analysis — p-value is for Diastolic BP change from baseline (Week 1) to Week 25; [statistical method as in outcome 1, analysis 1]

15. Secondary Outcome: Change From Baseline in Pulse Rate
Time Frame: baseline (Week 1), Week 13, Week 25
Population: All randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 246 | 118
beats per minute (bpm)
  Week 13 Change | 0.03 (0.60) | -1.56 (0.88)
  Week 25 Change | 2.10 (0.69) | -0.87 (1.28)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.121, Mixed Models Analysis — p-value is for change from baseline (Week 1) to Week 13; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.038, Mixed Models Analysis — p-value is for change from baseline (Week 1) to Week 25; [statistical method as in outcome 1, analysis 1]

16. Secondary Outcome: Change From Baseline in Weight
Time Frame: baseline (Week 1), Week 13, Week 25
Population: All randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 248 | 121
kilograms (kg)
  Week 13 Change | -0.86 (0.17) | 0.06 (0.26)
  Week 25 Change | -0.69 (0.22) | -0.03 (0.38)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — p-value is for Weight change from baseline (Week 1) to Week 13; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.127, Mixed Models Analysis — p-value is for Weight change from baseline (Week 1) to Week 25; [statistical method as in outcome 1, analysis 1]

17. Secondary Outcome: Number of Participants With Abnormal Vital Signs and Weight at Any Time During the Study
Description: A patient has a treatment-emergent elevated supine systolic blood pressure if the value is ≥140 with an increase ≥10 from baseline. A patient has a treatment-emergent elevated supine diastolic blood pressure if the value is ≥90 with an increase ≥10 from baseline. A patient has a treatment-emergent elevated supine pulse if the value is ≥100 with an increase ≥10 from baseline.
  A patient has abnormal weight change if the gain or loss is ≥7% compared to baseline.
Time Frame: Baseline (Week 1) through Week 25
Population: All randomized patients with a normal baseline and at least one post-baseline value in each treatment group.
Measure: Number; unit: Participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 248 | 121
Participants
  Diastolic Blood Pressure - High (n=210, n=98) | 22 | 5
  Pulse - High (n=243, n=115) | 10 | 4
  Systolic Blood Pressure - High (n=119, n=58) | 28 | 7
  Weight Change (gain) | 11 | 2
  Weight Change (loss) | 15 | 6
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.135, Fisher Exact — p-value is for Diastolic Blood Pressure
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Pulse; Test type: Superiority or Other; p = 1.00, Fisher Exact — p-value is for Pulse
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.107, Fisher Exact — p-value is for Systolic Blood Pressure
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.235, Fisher Exact — p-value is for Weight Change (gain)
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.813, Fisher Exact — p-value is for Weight Change (loss)

18. Secondary Outcome: Number of Participants Experiencing Sustained Hypertension (SH) or Orthostatic Hypotension (OH)
Description: Sustained Hypertension is defined as supine systolic BP >= 140 (or diastolic BP >= 90) mm Hg and increase from baseline (highest value in baseline visit interval) >= 10 mm Hg for 3 or more consecutive visits in postbaseline visit interval. Orthostatic Hypotension is defined as standing diastolic BP at least 10 mm Hg less than the supine diastolic BP or the standing systolic BP at least 20 mm Hg less than the supine systolic BP at any time in postbaseline visit interval and a patient does not meet this criterion at any visit in baseline interval.
Time Frame: baseline (Week 1) through Week 25
Population: All randomized patients with a normal baseline and at least one post-baseline value in each treatment group.
Measure: Number; unit: Participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 246 | 118
Participants
  Sustained Hypertension | 5 | 1
  Orthostatic Hypotension (n=183, n=90) | 57 | 21
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.668, Fisher Exact — p-value is for Sustained Hypertension
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.201, Fisher Exact — p-value is for Orthostatic Hypotension

19. Secondary Outcome: Summary of Adverse Events and Serious Adverse Events Leading to Discontinuation
Description: Adverse Events and Serious Adverse Events leading to study discontinuation.
Time Frame: baseline (Week 1) through Week 25
Population: All randomized patients.
Measure: Number; unit: participants
Groups:
- Placebo Non-rescue: Participants who were randomized to placebo at baseline and for whom treatment rescue was not required during continuation phase. Participants received placebo for 13 weeks (The first week was placebo lead-in). This double-blind acute phase was followed by a double-blind 12 week continuation phase during which they continued to receive placebo until completing or discontinuing from the study.
- Placebo Rescue: Participants who were randomized to placebo at baseline and for whom rescue treatment was required during the continuation phase. Participants received placebo for 13 weeks (The first week was placebo lead-in). This double-blind acute phase was followed by a double-blind 12 week continuation phase during which they were rescued to duloxetine 60 milligrams (mg) orally once daily (QD) beginning with duloxetine 30 mg QD orally for one week followed by duloxetine 60 mg QD orally until completing or discontinuing from the study.
Arm/Group | Duloxetine | Placebo Non-rescue | Placebo Rescue
Number analyzed (Participants) | 249 | 86 | 35
participants
  Total Discontinued due to Adverse Events | 38 | 7 | 0
  Diarrhoea | 3 | 0 | 0
  Fatigue | 3 | 0 | 0
  Headache | 1 | 2 | 0
  Nausea | 3 | 0 | 0
  Constipation | 2 | 0 | 0
  Dizziness | 2 | 0 | 0
  Hypertension | 1 | 1 | 0
  Memory impairment | 2 | 0 | 0
  Urinary Tract Infection | 2 | 0 | 0
  Vomiting | 1 | 1 | 0
  Alopecia | 1 | 0 | 0
  Anxiety | 1 | 0 | 0
  Blood pressure increased | 0 | 1 | 0
  Chills | 1 | 0 | 0
  Depression | 1 | 0 | 0
  Erectile dysfunction | 1 | 0 | 0
  Faecal incontinence | 1 | 0 | 0
  Gastrooesophageal reflux disease | 1 | 0 | 0
  Hip fracture | 1 | 0 | 0
  Insomnia | 1 | 0 | 0
  Intracranial aneurysm | 1 | 0 | 0
  Lethargy | 1 | 0 | 0
  Oesophageal adenocarcinoma metastatic | 1 | 0 | 0
  Palpitations | 1 | 0 | 0
  Paranasal sinus hypersecretion | 1 | 0 | 0
  Pneumoperitoneum | 1 | 0 | 0
  Presyncope | 0 | 1 | 0
  Rash pruritic | 0 | 1 | 0
  Renal failure acute | 1 | 0 | 0
  Suicidal ideation | 1 | 0 | 0
  Tremor | 1 | 0 | 0

20. Secondary Outcome: Change From Baseline in Laboratory Values - Platelet Count
Description: Results are reported for laboratory analytes that exhibited statistically significantly different changes from baseline to endpoint between treatment groups. Statistical significance was considered at the 0.05 level.
Time Frame: baseline (Week 1), Week 13, Week 25
Population: All randomized patients with a baseline and at least one post-baseline value in each treatment group.
Measure: Mean (Standard Deviation); unit: billions per liter (bill/L)
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 227 | 108
billions per liter (bill/L)
  Platelet Count Week 13 Change | 7.92 (45.75) | -4.66 (42.95)
  Platelet Count Week 25 Change | 10.58 (51.66) | -6.11 (39.87)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, ANOVA — p-value is for Platelet Count change from baseline (Week 1) to Week 13; Model: Change=Treatment+Pooled Investigator
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — p-value is for Platelet Count change from baseline (Week 1) to Week 25; Model: Change=Treatment+Pooled Investigator

21. Secondary Outcome: Change From Baseline in Laboratory Values - Uric Acid
Description: as for outcome 20
Time Frame: baseline (Week 1), Week 13, Week 25
Population: All randomized patients with a baseline and at least one post-baseline value in each treatment group.
Measure: Mean (Standard Deviation); unit: micromole/liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 230 | 112
micromole/liter
  Week 13 Change | -11.63 (63.05) | 9.30 (47.39)
  Week 25 Change | -9.93 (59.64) | 10.26 (48.29)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — p-value is for Uric Acid change from baseline (Week 1) to Week 13; Model: Change = Treatment + Pooled Investigator
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — p-value is for Uric Acid change from baseline (Week 1) to Week 25; Model: Change = Treatment + Pooled Investigator

22. Secondary Outcome: Change From Baseline in Laboratory Values - Erythrocyte Count
Description: as for outcome 20
Time Frame: baseline (Week 1), Week 25
Population: All randomized patients with a baseline and at least one post-baseline value in each treatment group.
Measure: Mean (Standard Deviation); unit: Trillion/Liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 228 | 109
Trillion/Liter
  Erythrocyte Count | -0.04 (0.29) | 0.01 (0.25)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.014, ANOVA — p-value is for Erythrocyte Count change from baseline (Week 1) to Week 25; Model: Change=Treatment+Pooled Investigator

23. Secondary Outcome: Change From Baseline in Laboratory Values - Hemoglobin, Mean Cell Hemoglobin Concentration (MCHC)
Description: as for outcome 20
Time Frame: baseline (Week 1), Week 25
Population: All randomized patients with a baseline and at least one post-baseline value in each treatment group.
Measure: Mean (Standard Deviation); unit: Micromole/liter (Fe)
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 228 | 109
Micromole/liter (Fe)
  Hemoglobin Week 25 Change | -0.11 (0.56) | 0.01 (0.46)
  Mean Cell Hemoglobin Concentration Week 25 Change | -0.20 (0.81) | -0.02 (0.81)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.019, ANOVA — p-value is for Hemoglobin change from baseline (Week 1) to Week 25; Model: Change = Treatment + Pooled Investigator
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.048, ANOVA — p-value is for Mean Cell Hemoglobin Concentration change from baseline (Week 1) to Week 25; Model: Change=Treatment+Pooled Investigator

24. Secondary Outcome: Change From Baseline in Laboratory Values - Chloride and Fasting Glucose
Description: as for outcome 20
Time Frame: baseline (Week 1), Week 25
Population: All randomized patients with a baseline and at least one post-baseline value in each treatment group.
Measure: Mean (Standard Deviation); unit: millimole/liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 230 | 112
millimole/liter
  Chloride Week 25 Change | -0.63 (2.83) | 0.01 (2.77)
  Fasting Glucose Week 25 Change (n=155, n=67) | 0.37 (1.88) | -0.11 (1.06)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.040, ANOVA — p-value is for Chloride change from baseline (Week 1) to Week 25; Model: Change = Treatment + Pooled Investigator
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.036, ANOVA — p-value is for Fasting Glucose change from baseline (Week 1) to Week 25; Model: Change=Treatment+Pooled Investigator

25. Secondary Outcome: Number of Participants With Abnormal Laboratory Values - Low Leukocyte Count
Description: The number of participants with abnormal laboratory values at any time during the study period. Results are reported for laboratory analytes that exhibited statistically significantly different proportions of participants who had abnormal values between treatment groups. Statistical significance was considered at the 0.05 level. The lower limit of normal for leukocyte count is 3.8 Billion/Liter. Participants who had a value below that number were considered to have abnormally low leukocyte count.
Time Frame: baseline (Week 1) through Week 13
Population: All randomized patients with a normal baseline and at least one post-baseline value in each treatment group.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 225 | 109
participants
  Leukocyte Count (Low) | 11 | 0
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.019, Fisher Exact

26. Secondary Outcome: Change From Baseline in Electrocardiograms
Description: The Electrocardiogram measures include the following time intervals: QT interval, QT Interval Corrected for Heart Rate Using Fridericia's Formula (QTcF), QT Interval Corrected for Heart Rate Using Bazett's Formula (QTcB), PR interval and QRS interval.
Time Frame: baseline (Week 1), Week 25
Population: Participants with a baseline and at least one non-missing post baseline value.
Measure: Least Squares Mean (Standard Error); unit: millisecond (msec)
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 194 | 68
millisecond (msec)
  QT Interval Week 25 Change | -11.80 (2.19) | -10.95 (3.43)
  QTcF Interval Week 25 Change | -5.02 (1.48) | -5.91 (2.33)
  QTcB Interval Week 25 Change | -1.38 (1.61) | -3.78 (2.55)
  PR Interval Week 25 Change | -5.91 (1.45) | -1.34 (2.32)
  QRS Interval Week 25 Change | -1.11 (0.80) | -3.25 (1.26)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.815, ANCOVA — p-value is for QT Interval change from baseline (Week 1) to Week 25; Model: Change=Treatment+Pooled Investigator+Baseline
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.721, ANCOVA — p-value is for QTcF Interval change from baseline (Week 1) to Week 25; Model: Change=Treatment+Pooled Investigator+Baseline
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.376, ANCOVA — p-value is for QTcB Interval change from baseline (Week 1) to Week 25; Model: Change=Treatment+Pooled Investigator+Baseline
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.065, ANCOVA — p-value is for PR Interval change from baseline (Week 1) to Week 25; Model: Change=Treatment+Pooled Investigator+Baseline
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.110, ANCOVA — p-value is for QRS Interval change from baseline (Week 1) to Week 25; Model: Change=Treatment+Pooled Investigator+Baseline

27. Secondary Outcome: Number of Participants With Successful Treatment Outcome
Description: Successful treatment outcome defined as: Participant completed the study and being in remission (HAMD-17 Total score ≤7 and ≤10) at least for the last two visits (4 weeks)of the study. The HAMD-17 is used to assess the severity of depression. The total score ranges from 0 (not at all depressed) to 52 (severely depressed).
Time Frame: Baseline (Week 1) through Week 25
Population: All participants randomized under protocol amendment c,d,e, and that have non-missing successful treatment values.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 204 | 95
participants
  Successful Treatment Outcome (with HAMD17 ≤ 7) | 55 | 17
  Successful Treatment Outcome (with HAMD17 ≤ 10) | 74 | 21
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.110, Fisher Exact — p-value is for Successful Treatment Outcome defined with HAMD-17 ≤7 criteria
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.016, Fisher Exact — p-value is for Successful Treatment Outcome defined with HAMD-17 ≤10 criteria

28. Secondary Outcome: Change From Baseline on Cognitive Test Scores: Verbal Learning and Recall Test (VLRT), Symbol Digit Substitution Test (SDST), Trail Making Test (Part B), 2-Digit Cancellation Test (2DCT), and the Composite Cognitive Score Derived From the Above Scores
Description: The cognitive assessment battery is composed of four tests: Verbal Learning (score 0-15)and Delayed Recall(score 0-15) test, SDST(Score 0-133),2DCT(score 0-40),Trail Making(Part B)(score 0-180).They are designed to challenge the patient's abilities in the following areas: verbal learning and memory; attention to visually presented material; and working memory and executive function. Composite Cognitive score(0-51)is derived from normalized individual test scores. For Trail Making Test,lower number indicates better cognition. For all other test scores,higher number indicates better cognition.
Time Frame: baseline (Week 1), Week 9, Week 25
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 183 | 90
units on a scale
  Composite Cognitive Score Week 9 | -0.38 (0.38) | 0.01 (0.51)
  Composite Cognitive Score Week 25 | 0.96 (0.40) | 0.31 (0.54)
  Learning Trials Score Week 9 | -0.06 (0.12) | -0.04 (0.17)
  Learning Trials Score Week 25 | 0.34 (0.13) | 0.06 (0.18)
  Delayed Recall Score Week 9 | -0.65 (0.21) | -0.59 (0.28)
  Delayed Recall Score Week 25 | 0.12 (0.22) | -0.36 (0.29)
  SDST Score Week 9 | 1.98 (0.76) | 3.99 (1.04)
  SDST Score Week 25 | 5.60 (0.84) | 3.61 (1.15)
  2DCT Score Week 9 | 0.30 (0.46) | 0.94 (0.63)
  2DCT Score Week 25 | 0.87 (0.51) | 1.01 (0.70)
  Trail Making Test (Part B) Week 9 | -5.60 (2.90) | -3.09 (4.00)
  Trail Making Test (Part B) Week 25 | -1.59 (2.82) | -6.86 (3.86)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.511, ANCOVA — p-value is for Composite Cognitive Score change from baseline (Week 1) to Week 9; Model: Change=Treatment+Pooled Investigator+Baseline
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.300, ANCOVA — p-value is for Composite Cognitive Score change from baseline (Week 1) to Week 25; Model: Change=Treatment+Pooled Investigator+Baseline
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.922, ANCOVA — p-value is for Learning Trials Score change from baseline (Week 1) to Week 9; Model: Change=Treatment+Pooled Investigator+Baseline
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.190, ANCOVA — p-value is for Learning Trials Score change from baseline (Week 1) to Week 25; Model: Change=Treatment+Pooled Investigator+Baseline
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.850, ANCOVA — p-value is for Delayed Recall Score change from baseline (Week 1) to Week 9; Model: Change=Treatment+Pooled Investigator+Baseline
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.158, ANCOVA — p-value is for Delayed Recall Score change from baseline (Week 1) to Week 25; Model: Change=Treatment+Pooled Investigator+Baseline
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.099, ANCOVA — p-value is for SDST Score change from baseline (Week 1) to Week 9; Model: Change=Treatment+Pooled Investigator+Baseline
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.141, ANCOVA — p-value is for SDST Score change from baseline (Week 1) to Week 25; Model: Change=Treatment+Pooled Investigator+Baseline
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.379, ANCOVA — p-value is for 2DCT Score change from baseline (Week 1) to Week 9; Model: Change=Treatment+Pooled Investigator+Baseline
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.858, ANCOVA — p-value is for 2DCT Score change from baseline (Week 1) to Week 25; Model: Change=Treatment+Pooled Investigator+Baseline
Statistical Analysis 11: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.591, ANCOVA — p-value is for Trail Making Test Score change from baseline (Week 1) to Week 9; Model: Change=Treatment+Pooled Investigator+Baseline
Statistical Analysis 12: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.242, ANCOVA — p-value is for Trail Making Test Score change from baseline (Week 1) to Week 25; Model: Change=Treatment+Pooled Investigator+Baseline

ADVERSE EVENTS:
Time Frame: Baseline (Week 1) through Week 25.
Description: The event of fall was collected using a solicited Falls Assessment questionnaire at each visit.
Groups:
- Placebo: Participants received placebo for 13 weeks (The first week was placebo lead-in). This double-blind acute phase was followed by a double-blind 12 week continuation phase during which participants either remained on placebo or were eligible for receiving duloxetine 60 milligrams (mg) orally once daily (QD), beginning with duloxetine 30 mg QD orally for 1 week followed by duloxetine 60 mg QD orally for the remainder of the study based on depression symptom severity. Results are for the randomized placebo patients who reported events while they were on placebo.
- Rescued Placebo: Participants received placebo for 13 weeks (The first week was placebo lead-in). This double-blind acute phase was followed by a double-blind 12 week continuation phase during which participants were rescued to duloxetine 60 milligrams (mg) orally once daily (QD) beginning with duloxetine 30 mg QD orally for one week followed by duloxetine 60 mg QD orally for the remainder of the study. Results are for the randomized placebo patients who were rescued to duloxetine and reported events while they were on duloxetine.
Arm/Group | Duloxetine | Placebo | Rescued Placebo
Serious Adverse Events (participants affected / at risk) | 13/249 | 4/121 | 1/35
Other Adverse Events (participants affected / at risk) | 199/249 | 77/121 | 17/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=249) | Placebo (N=121) | Rescued Placebo (N=35)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Abscess intestinal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toe amputation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=249) | Placebo (N=121) | Rescued Placebo (N=35)
Constipation (Gastrointestinal disorders) | 37 (37) | 5 (6) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 31 (33) | 3 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 34 (35) | 7 (7) | 1 (1)
Nausea (Gastrointestinal disorders) | 28 (29) | 7 (7) | 0 (0)
Fatigue (General disorders) | 14 (17) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 13 (14) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 12 (16) | 4 (4) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 59 (80) | 17 (21) | 6 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (14) | 8 (9) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (11) | 2 (3) | 2 (2)
Dizziness (Nervous system disorders) | 26 (30) | 6 (7) | 2 (2)
Headache (Nervous system disorders) | 32 (37) | 13 (13) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 15 (15) | 2 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 5 (5) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days